CLINICAL TRIAL: NCT05751837
Title: Feasibility Study of Intra-Tumoral Lipopolysaccharide Immunotherapy for Intra-Abdominal
Acronym: LPS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Patrick Wagner, MD, FACS (Other)
Collaborators: List Biological Laboratories, Inc (Unknown)
Responsible Party: Sponsor-Investigator, Patrick Wagner, MD, FACS, Director, AHNCI Division of Complex General Surgical Oncology, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-263
Record Dates: First submitted 2023-02-02; First posted 2023-03-02 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-07

CONDITIONS: Abdominal Cancer; Malignancy
MeSH Terms: conditions — Neoplasms | interventions — Lipopolysaccharides

STUDY DESIGN:
Intervention Model Description: Single-arm, open label, comparative, phase I safety and feasibility study, with correlative translational studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm (Experimental): Injection of Lipopolysaccharide into one abdominal tumor
  Interventions: Biological: Lipopolysaccharide

INTERVENTIONS:
Biological: Lipopolysaccharide — One tumor will be injected with 1 ug LPS (investigational drug) over approximately one minute
  Other Names: LPS; E. coli 0113

SUMMARY:
The purpose of this research study is to determine whether a sterile bacteria wall chemical, called lipopolysaccharide (LPS), can be injected safely into abdominal tumors during routine laparoscopic surgery performed as a preliminary procedure in patients who will subsequently undergo a larger planned operation to remove abdominal tumors. The researchers will biopsy the tumor before injection and then again at the time of the larger operation to assess whether any effect of the treatment can be measured.

DETAILED DESCRIPTION:
Immunotherapy for advanced cancers of the abdomen can be quite effective, but not all tumors are responsive to this type of treatment. There is intense interest in new methods to convert non-responsive tumors into responsive tumors. One such method is to inject chemical constituents of micro-organisms into tumors in order to stimulate the immune system to recognize the tumor as foreign and mount an immune response to treatment.

Provide a concise and brief, one-paragraph summary of your research project. Include a summary of the problem, the main objective and rationale of your project; a brief description of the experimental approach and methods; a concise description/summary of the most important results that you hope to obtain; and why think your results will be significant

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 to 99 years
2. Pre-menopausal women less than or equal to18 years of age must have a negative urine/serum pregnancy test prior to standard-of-care surgery and investigational treatment.
3. Participants must have an advanced intra-abdominal tumor, including metastatic or recurrent, biopsy-proven, digestive tract tumors.
4. Participants must have at least two index non-visceral intra-abdominal tumors that are grossly visible, >1cm3 in volume, and amenable to biopsy and injection of investigational drug or control solution at the time of laparoscopy.
5. Participants must be planning or scheduled to undergo a standard-of-care abdominal laparoscopic surgical procedure at AGH or WPH and be potentially eligible for a second, definitive operation to remove the tumor(s) pending the findings during laparoscopy.
6. Must be able to read and understand English and consent for themselves

Exclusion Criteria:

1. Pregnant or lactating females
2. Investigational drug use within 30 days prior to enrollment.
3. Immunosuppressive medication including corticosteroids within 30 days prior to enrollment.
4. Active chemotherapy or radiotherapy within 4 weeks of investigational agent injection.
5. Active infection requiring systemic therapy or causing fever >38.1 degree C or unexplained fever >38.1 degree C within seven days prior to investigational agent injection
6. Laboratory abnormalities, drawn according to standard clinical care in anticipation of upcoming surgery outside the following limits:

   AST/SGOT > 1.5 times the upper limit of normal ALT/SGPT > 1.5 times the upper limit of normal Total bilirubin > 1.5 times the upper limit of normal Creatinine > 1.5 times the upper limit of normal Hemoglobin < 9 gm/dL White blood cell count < 3,000/ mm3 Platelet count < 70,000/mm3 INR >1.5 times the upper limit of normal PTT >1.5 times the upper limit of normal
7. History of allergic reaction to the investigational agent carrier solution.
8. Medical contra-indication or allergic reaction to acetaminophen or NSAIDs.
9. Participants who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
10. Adverse events from prior therapy that have not resolved to CTCAE version 5 grade < and equal to1 prior to enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 30 Days
  The number, nature and severity of adverse events as assessed by CTCAE v 4.0 will be determined in a series of six patients undergoing injection of bacterial-derived immunotherapeutic toll receptor agonist (LPS) instilled via direct injection into intra-abdominal tumors during laparoscopic surgery.

SECONDARY OUTCOMES:
Alteration in Cellular and Soluble Immune Biomarkers in Injected Tumors | 30 days
  Changes in intra-tumoral leukocyte subgroup densities and soluble immune biomarker concentrations will be assessed in injected tumors and compared against non-injected tumors.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Allegheny Health Network Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Allegheny Health Network West Penn Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be used for future study without first obtaining IRB approval. The investigator will obtain a data use agreement between the provider (the PI) of the data and any recipient researchers before sharing data.

REFERENCES:
- [Background] Shetab Boushehri MA, Lamprecht A. TLR4-Based Immunotherapeutics in Cancer: A Review of the Achievements and Shortcomings. Mol Pharm. 2018 Nov 5;15(11):4777-4800. doi: 10.1021/acs.molpharmaceut.8b00691. Epub 2018 Oct 3. PMID 30226786
- [Background] Oblak A, Jerala R. Toll-like receptor 4 activation in cancer progression and therapy. Clin Dev Immunol. 2011;2011:609579. doi: 10.1155/2011/609579. Epub 2011 Nov 3. PMID 22110526
- [Background] Berendt MJ, North RJ, Kirstein DP. The immunological basis of endotoxin-induced tumor regression. Requirement for a pre-existing state of concomitant anti-tumor immunity. J Exp Med. 1978 Dec 1;148(6):1560-9. doi: 10.1084/jem.148.6.1560. PMID 309922
- [Background] Chicoine MR, Won EK, Zahner MC. Intratumoral injection of lipopolysaccharide causes regression of subcutaneously implanted mouse glioblastoma multiforme. Neurosurgery. 2001 Mar;48(3):607-14; discussion 614-5. doi: 10.1097/00006123-200103000-00032. PMID 11270552
- [Background] Mariani CL, Rajon D, Bova FJ, Streit WJ. Nonspecific immunotherapy with intratumoral lipopolysaccharide and zymosan A but not GM-CSF leads to an effective anti-tumor response in subcutaneous RG-2 gliomas. J Neurooncol. 2007 Dec;85(3):231-40. doi: 10.1007/s11060-007-9415-2. Epub 2007 Jun 14. PMID 17568998
- [Background] Goto S, Sakai S, Kera J, Suma Y, Soma GI, Takeuchi S. Intradermal administration of lipopolysaccharide in treatment of human cancer. Cancer Immunol Immunother. 1996 May;42(4):255-61. doi: 10.1007/s002620050279. PMID 8665574
- [Background] Engelhardt R, Mackensen A, Galanos C. Phase I trial of intravenously administered endotoxin (Salmonella abortus equi) in cancer patients. Cancer Res. 1991 May 15;51(10):2524-30. PMID 2021932
- [Background] van Lier D, Geven C, Leijte GP, Pickkers P. Experimental human endotoxemia as a model of systemic inflammation. Biochimie. 2019 Apr;159:99-106. doi: 10.1016/j.biochi.2018.06.014. Epub 2018 Jun 22. PMID 29936295
- [Background] Fong YM, Marano MA, Moldawer LL, Wei H, Calvano SE, Kenney JS, Allison AC, Cerami A, Shires GT, Lowry SF. The acute splanchnic and peripheral tissue metabolic response to endotoxin in humans. J Clin Invest. 1990 Jun;85(6):1896-904. doi: 10.1172/JCI114651. PMID 2347917
- [Background] Calvano SE, Coyle SM. Experimental human endotoxemia: a model of the systemic inflammatory response syndrome? Surg Infect (Larchmt). 2012 Oct;13(5):293-9. doi: 10.1089/sur.2012.155. Epub 2012 Oct 16. PMID 23072275
- [Background] Vila G, Riedl M, Resl M, van der Lely AJ, Hofland LJ, Clodi M, Luger A. Systemic administration of oxytocin reduces basal and lipopolysaccharide-induced ghrelin levels in healthy men. J Endocrinol. 2009 Oct;203(1):175-9. doi: 10.1677/JOE-09-0227. Epub 2009 Jul 8. PMID 19587265
- [Background] Hudgins LC, Parker TS, Levine DM, Gordon BR, Saal SD, Jiang XC, Seidman CE, Tremaroli JD, Lai J, Rubin AL. A single intravenous dose of endotoxin rapidly alters serum lipoproteins and lipid transfer proteins in normal volunteers. J Lipid Res. 2003 Aug;44(8):1489-98. doi: 10.1194/jlr.M200440-JLR200. Epub 2003 May 16. PMID 12754273
- [Background] Mehta RS, Nishihara R, Cao Y, Song M, Mima K, Qian ZR, Nowak JA, Kosumi K, Hamada T, Masugi Y, Bullman S, Drew DA, Kostic AD, Fung TT, Garrett WS, Huttenhower C, Wu K, Meyerhardt JA, Zhang X, Willett WC, Giovannucci EL, Fuchs CS, Chan AT, Ogino S. Association of Dietary Patterns With Risk of Colorectal Cancer Subtypes Classified by Fusobacterium nucleatum in Tumor Tissue. JAMA Oncol. 2017 Jul 1;3(7):921-927. doi: 10.1001/jamaoncol.2016.6374. PMID 28125762
- [Background] Kiers D, Leijte GP, Gerretsen J, Zwaag J, Kox M, Pickkers P. Comparison of different lots of endotoxin and evaluation of in vivo potency over time in the experimental human endotoxemia model. Innate Immun. 2019 Jan;25(1):34-45. doi: 10.1177/1753425918819754. PMID 30782041
- [Background] Coley WB. II. Contribution to the Knowledge of Sarcoma. Ann Surg. 1891 Sep;14(3):199-220. doi: 10.1097/00000658-189112000-00015. No abstract available. PMID 17859590
- [Background] Coley WB. The treatment of malignant tumors by repeated inoculations of erysipelas. With a report of ten original cases. 1893. Clin Orthop Relat Res. 1991 Jan;(262):3-11. No abstract available. PMID 1984929
- [Background] Otto F, Schmid P, Mackensen A, Wehr U, Seiz A, Braun M, Galanos C, Mertelsmann R, Engelhardt R. Phase II trial of intravenous endotoxin in patients with colorectal and non-small cell lung cancer. Eur J Cancer. 1996 Sep;32A(10):1712-8. doi: 10.1016/0959-8049(96)00186-4. PMID 8983279
- [Background] Millischer V, Heinzl M, Faka A, Resl M, Trepci A, Klammer C, Egger M, Dieplinger B, Clodi M, Schwieler L. Intravenous administration of LPS activates the kynurenine pathway in healthy male human subjects: a prospective placebo-controlled cross-over trial. J Neuroinflammation. 2021 Jul 17;18(1):158. doi: 10.1186/s12974-021-02196-x. PMID 34273987
- [Background] Humeau J, Le Naour J, Galluzzi L, Kroemer G, Pol JG. Trial watch: intratumoral immunotherapy. Oncoimmunology. 2021 Oct 15;10(1):1984677. doi: 10.1080/2162402X.2021.1984677. eCollection 2021. PMID 34676147